CLINICAL TRIAL: NCT01536223
Title: Cisplatin and 5-fluorouracil(PF) or Docetaxel,Cisplatin and 5-fluorouracil (TPF) Neoadjuvant Chemotherapy With Chemoradiation Therapy for Locally Advanced Nasopharyngeal Carcinoma--A Randomised Prospective Multicenter Phase 3 Study
Brief Title: Efficacy Study of Neoadjuvant Chemotherapy With Chemoradiation Therapy for Nasopharyngeal Carcinoma
Acronym: ESNCCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang University (Other); Zhejiang Provincial People's Hospital (Other); Sir Run Run Shaw Hospital (Other); Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH13
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2012-04

CONDITIONS: Chemoradiation; Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma (NPC); cisplatin and 5-fluorouracil (PF); docetaxel,cisplatin and 5-fluorouracil(TPF); Neoadjuvant Chemotherapy; intensity modulated radiotherapy(IMRT)
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Fluorouracil; Population Groups; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF group (Active Comparator): the group of participants who undergoing cisplatin and 5-fluorouracil(PF)neoadjuvant chemotherapy
  Interventions: Drug: PF (cisplatin and 5-fluorouracil) group
- TPF group (Experimental): TPF(docetaxel , cisplatin and 5-fluorouracil)neoadjuvant chemotherapy
  Interventions: Drug: TPF (docetaxel plus cisplatin and 5-fluorouracil) group

INTERVENTIONS:
Drug: PF (cisplatin and 5-fluorouracil) group — the group the patients using PF(cisplatin and 5-fluorouracil )neoadjuvant chemotherapy 3 cycles of neoadjuvant chemotherapy at day1,22 and 43 with cisplatin 100mg/m2 and 5-fluorouracil 4000mg/m2 civ 120 hours And then chemoradiation using IMRT with 2 cycles of cisplatin concurrent chemotherapy at 80mg/m2.
  Other Names: Active Comparator group
  Arms: PF group
Drug: TPF (docetaxel plus cisplatin and 5-fluorouracil) group — 3 cycles of TPF neoadjuvant chemotherapy at day1,22 and 43 with docetaxel 75mg/m2,cisplatin75mg/m2 and 5-fluorouracil 2400mg/m2 civ 96 hours .
  And then chemoradiation using IMRT with 2 cycles of cisplatin concurrent chemotherapy at 80mg/m2.
  Other Names: Experiment group
  Arms: TPF group

SUMMARY:
Locally advanced nasopharyngeal carcinoma patients(UICC7th stageIII to IVb) will receive either cisplatin plus 5-fluorouracil (PF) or docetaxel plus cisplatin and 5-fluorouracil(TPF) neoadjuvant chemotherapy with concurrent chemoradiation.

DETAILED DESCRIPTION:
For locally advanced nasopharyngeal carcinoma patients(UICC7th stageIII to IVb),the investigators randomised assign to either 3 cycles of cisplatin plus 5-fluorouracil plus (PF) or 3 cycles of docetaxel plus cisplatin and 5-fluorouracil(TPF) neoadjuvant chemotherapy. 21 days a cycle.

After the neoadjuvant chemotherapy ,the patients will receive the intensity modulated radiotherapy(IMRT) with 2 cycles of concurrent chemotherapy of cisplatin 80mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing carcinoma.
2. Tumor staged as N2-3 or T3-4N1(according to the 7th AJCC staging system)
3. No evidence of distant metastasis(M0)
4. Performance status:KPS>70
5. With normal liver function test(ALT, AST<1.5ULN)
6. Renal:creatinine clearance >60ml/min
7. Without hematopathy,marrow:WBC>4*109/L, HGB>80G/L, and PLT>100*109/L.
8. With controled blood glucose for diabetes patients
9. Written informed consent

Exclusion Criteria:

1. WHO type I squamous cell carcinoma or adenocarcinoma
2. Age>70 or <18
3. With a history of renal disease
4. Prior malignancy (except adequately treated carcinoma in-situ of the cervix or basal/squamous cell carcinoma of the skin0
5. Previous chemotherapy or radiotherapy(except non-melanomatous skin cancers outside the intended RT treatment volume)
6. Patient is pregnant or lactating .
7. Peripheral neuropathy
8. Emotional disturbance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
3-year progress free survival(PFS) | 3 years after the inception assignment
  PFS means assignment to the date of any local or distant progress of the disease using Kaplan-Meier calculate the progress free survival rates,and find out is there significant difference between these two groups.

SECONDARY OUTCOMES:
overall survival(OS) | 2 years ,3 years and 5 years after the inception of the assignment
  the overall survival denote to assignment to date of death from any cause. Using Kaplan-Meier to calculate the 2-year ,3-year,5-year overall survival rate,and find is there any significant difference between these two groups.
Adverse events | participants will be followed for the duration of hospital stay,an expected average of 100 days and every 3 months thereafter for 5 years
  observe and record the toxicity profile(including but not limit to mucositis,liver and kidney function,et al.)according NCI-CTCAE(3rd edition) during the neoadjuvant chemotherapy ,chemoradiation and follow-up.
local control rate (LCR) | 1 year ,2 years,3 years and 5 years after the inception of the study

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Jin T, Qin WF, Jiang F, Jin QF, Wei QC, Jia YS, Sun XN, Li WF, Chen XZ. Cisplatin and Fluorouracil Induction Chemotherapy With or Without Docetaxel in Locoregionally Advanced Nasopharyngeal Carcinoma. Transl Oncol. 2019 Apr;12(4):633-639. doi: 10.1016/j.tranon.2019.01.002. Epub 2019 Feb 20. PMID 30797141